CLINICAL TRIAL: NCT00381602
Title: A Phase II, Randomized, Cross-Over, Vehicle-Controlled, Double-Blind, Multicenter Study of the Safety, Pharmacodynamics, and Preliminary Efficacy of GHRP-1/AG in Subjects With ESRD on Hemodialysis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrolment
Sponsor: QLT Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GHRP ESRD 01
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-03

CONDITIONS: End Stage Renal Disease
Keywords: End stage renal disease; Hemodialysis; Malnutrition; End stage renal disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic; Malnutrition

INTERVENTIONS:
Drug: GHRP-1/AG 70 mg depot in ESRD
Other: Placebo

SUMMARY:
Malnutrition and altered protein catabolism are serious problems in renal failure and hemodialysis (HD) patients. The purpose of this study is to characterize the safety of GHRP-1/AG in subjects with ESRD on HD; to characterize the pharmacodynamics (PD) of GHRP-1/AG in subjects with ESRD on HD by following GH and IGF-1; to describe the relationship between GHRP-1 PD and plasma concentrations of GHRP-1 and des-Ala-GHRP-1; and to evaluate the preliminary efficacy of GHRP-1/AG on nutritional status of subjects with ESRD on HD using subjective global assessment of malnutrition inflammation scores (MIS) and changes in caloric intake.

DETAILED DESCRIPTION:
This is a randomized, cross-over, double-blind, vehicle-controlled study. Subjects will receive single subcutaneous injections of the active GHRP-1/AG study treatment and vehicle control (ATRIGEL delivery system) in a randomized sequence. Each injection will be followed by a 4-week period of treatment exposure and a 2-week period of washout/follow-up. Treatments will be administered on the 2nd dialysis day of a 3x/week dialysis schedule. The total duration of study participation will be 12 weeks. Safety will be followed throughtout the study with vital signs, electrocardiogram, clinical chemistry and hematology parameters, endocrine parameters, adverse events, and concomitant medications. PD effects of GHRP-1/AG will be evaluated by measuring GH, ICF-1, IGF-BP3, prolactin, and cortisol. Efficacy will be evaluated throughout the study with MIS, caloric intake, nPCR, dry weight, BMI, and albumin, BUN, creatinine, calcium, potassium, HGB, HCT, and CBC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ESRD who have been on HD for at least 3 months and have a urea reduction rate (URR) of at least 65%.
* Subjects who are 18 to 70 years of age.
* Subjects who have a body mass index (BMI) less than 30, albumin greater than 3.3 g/dL, and MIS of 5 to 10 (inclusive).

Exclusion Criteria:

* Subjects who have diabetes and are currently taking insulin.
* Subjects who have a history of or current significant central nervous system (CNS) disorders.
* Subjects who have active infection at baseline.
* Subjects who have active or unstable cardiac or arterial disease.
* Subjects who have uncontrolled tertiary hyperparathyroid condition.
* Subjects who have anemia.
* Subjects who have a history of hepatitis or current liver disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Vital signs
ECG
clinical chemistry and hematology
MIS
caloric intake (protein, fat, carbohydrates, total)
nPCR
BMI and dry weight
clinical laboratory parameters

SECONDARY OUTCOMES:
IGF-1, IGF-BP3, GH, prolactin, and cortisol plasma concentrations
GHRP-1 and des-Ala-GHRP-1 plasma concentrations
adverse events
concomitant medications
endocrine parameters

CONTACTS AND LOCATIONS:
Overall Officials: Graeme R Boniface, Study Director — QLT Inc.
Locations (2):
- United States (2):
  - Tulane University Medical School, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota